CLINICAL TRIAL: NCT07138443
Title: Influence of Melatonin on Cardiovascular and Skin Temperature Responses to Stress: A Randomized Controlled Trial
Brief Title: Influence of Melatonin on Cardiovascular and Thermoregulatory Responses to Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2241833-5
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stress; Mental Stress
Keywords: Melatonin; Mental stress; Trier Social Stress Test; Cardiovascular; Skin temperature
MeSH Terms: conditions — Stress, Psychological | interventions — Melatonin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the investigator and the participants will be blinded as to the condition that participants are in. A lab member who will be recused from data analysis and outcomes assessment will monitor participant assignment to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (3mg) (Experimental): Participants will ingest an acute oral melatonin tablet (3mg) prior to stress reactivity assessment.
  Interventions: Dietary Supplement: Melatonin 3 MG Oral Tablet
- Placebo (Placebo Comparator): Participants will ingest a placebo pill of the same color and shape as the melatonin tablet prior to reactivity assessment.
  Interventions: Dietary Supplement: Placebo Oral Tablet

INTERVENTIONS:
Dietary Supplement: Melatonin 3 MG Oral Tablet — Participants will ingest an acute 3mg oral melatonin tablet
  Arms: Melatonin (3mg)
Dietary Supplement: Placebo Oral Tablet — Participants will ingest a placebo tablet (sugar pill) of the same size, shape, and color of the active melatonin supplement
  Arms: Placebo

SUMMARY:
This study aims to evaluate the influence of acute oral melatonin supplementation on cardiovascular and skin temperature responses to mental stress. The hypothesis is that acute melatonin will lead to reduced cardiovascular and skin temperature responsiveness to acute mental stress.

DETAILED DESCRIPTION:
This study will utilize a randomized, crossover, placebo controlled experimental approach to determine the effects of acute oral melatonin supplementation (3mg) on blood pressure, heart rate, and regionalized skin temperature responsiveness to mental stress. The study will assess beat-by-beat blood pressure (finger plethysmography), continuous heart rate (electrocardiogram), and proximal/distal skin temperature continuously at rest and in response to the Trier Social Stress Test following either afternoon melatonin or placebo ingestion in a randomized order. Participants will consist of young healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18-70 years old.
* All subjects will be required to abstain from exercise and caffeine for 12 h, and alcohol for 24 h prior to the experiment.
* BMI must be <30 kg/m2.
* Menstruating women will initially be tested during their early follicular phase (2-5 days after initiating menstruation) or during low hormone phase (2-5 days after initiating menstruation) if on oral contraceptives to control for potential impact of sex steroids. Post-menopausal females (>5 years) will also be included. Females must have an intact uterus and at least one ovary. Use of hormonal replacement therapy will be allowed.

Exclusion Criteria:

* Circadian rhythm sleep disorders
* High obstructive sleep apnea diagnosis determined by STOP-BANG.
* History of meeting Diagnostic and Statistical Manual of Mental health (DSM-V) criteria of major psychiatric disorder
* Unstable or serious medical conditions (heart failure, diabetes, cardiovascular disease, etc.)
* Current, or use within past month, of psychoactive (other than stable treatment with antidepressant), hypnotic, stimulant or analgesic medication (except occasional non-narcotic analgesics), beta blockers, or alpha blockers
* Shift work or other types of self-imposed irregular sleep schedules
* Habitual smoking (6 or more cigarettes per week)
* Habitual alcohol consumption (more than 2 alcoholic drinks per day)
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Reactivity | 4 weeks
  Heart rate will be continuously monitored using electrocardiogram during a 10-minute baseline and in response to the Trier Social Stress Test. Heart rate reactivity during the stress will be quantified.
Blood Pressure Reactivity | 4 weeks
  Beat-by-beat systolic, diastolic, and mean arterial pressure will be assessed using finger plethysmography in response to the Trier Social Stress Test. Reactivity scores will be assessed by determining the difference in blood pressure during the stress task relative to baseline.
Distal-to-Proximal Skin Temperature Gradient | 4 weeks
  Skin temperature will be monitored using small temperature sensors (iButtons, type DS1922L; iButtonLink LLC) adhered to various distal and proximal regions of the body. Upper distal to proximal skin temperature gradients (DPG) will be calculated as the average skin temperature taken from the hand subtracted from the average skin temperature taken from the forearm/shoulder. Lower DPG will be calculated as the average skin temperature taken from the feet subtracted from the average skin temperature recorded at the calves.

SECONDARY OUTCOMES:
Perceived Stress and Coping (Likert Scale) | 4 weeks
  Participants' stress and perceived coping will be monitored throughout the stress task in both experimental conditions. Participants will be asked to rate their perceived stress on a Likert scale ranging from 1 (not at all stressed) to 7 (extremely stressed). Participants will also be asked to rate how well they perceived their ability to cope with the demands of the tasks on a scale ranging from 1 (not at all able to cope) to 7 (extremely able to cope). The quotient of stress/coping will be operationalized as a measure of threat perception. A challenge appraisal is defined as a stress-coping ratio of ≤1 (i.e., coping ability meets or exceeds the perceived stress of the task) whereas a threat appraisal is defined as a stress-coping ratio > 1 (i.e., perceived stress of the task exceeds coping abilities). Comparisons between conditions will be performed to assess the differences in numeric ratings of stress, coping, and threat perception measured in arbitrary units.
Karolinska Sleepiness Scale | 4 weeks
  The Karolinska Sleepiness Scale will be used to assess participants' reported sleepiness prior to stress task initiation. The scale ranges from 1 (extremely alert) to 10 (Extremely sleepy, can't stay awake) to measure momentary levels of sleepiness.
Salivary Melatonin | 4 weeks
  Saliva will be sampled 45 minutes after melatonin or placebo ingestion. This will be used to quantify salivary melatonin between conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Autonomic Function Laboratory, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No